CLINICAL TRIAL: NCT07310823
Title: IMMEDIATE AND SHORT-TERM EFFECT OF COMBINING SUBOCCIPITAL MYOFASCIAL RELEASE WITH MAITLAND MOBILIZATION ON CERVICOGENIC HEADACHE
Brief Title: Mangement of Cervicogenic Headache by Maual Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Alaa Mahmoud Ahmed, Msc candidate, orthopedic physical therapy department , cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CGH mangment
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cervicogenic Headache; Neck Pain Musculoskeletal
Keywords: cervicogenic headache; suboccipital myofacial release; maitland mobilization; neck pain; CROM
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial in which patients will be randomly assigned into three equal groups (19 patients per group) via the RANDOM.ORG method. Each group will receive a specific physical therapy management according the following:
  * Group A (Suboccipital Myofascial Release): Patients in this group will receive suboccipital myofascial release therapy for one session.
  * Group B (Maitland Mobilization): Patients in this group will receive Maitland mobilization therapy for one session.
  * Group C (Combined Group): Patients in this group will receive both techniques; suboccipital myofascial release therapy then Maitland mobilization for one session.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Suboccipital Myofascial Release) (Active Comparator): Patients in this group will receive suboccipital myofascial release therapy for one session.
  Interventions: Other: suboccipital myofacial release
- Group B (Maitland Mobilization) (Active Comparator): Patients in this group will receive Maitland mobilization therapy for one session.
  Interventions: Other: maitland mobilization
- Group C (Combined Group) (Active Comparator): Patients in this group will receive both techniques; suboccipital myofascial release therapy then Maitland mobilization for one session.
  Interventions: Other: combined myofacsial release with maitland mobilization

INTERVENTIONS:
Other: suboccipital myofacial release — one session of myofacial release for suboccipital muscle
  Arms: Group A (Suboccipital Myofascial Release)
Other: maitland mobilization — one session of upper cervical vertebral grade one and two mobilization
  Arms: Group B (Maitland Mobilization)
Other: combined myofacsial release with maitland mobilization — one session of myofacsial release and maitland mobilization for upper cervical and suboccipital muscle
  Arms: Group C (Combined Group)

SUMMARY:
This study aims to investigate immediate and short-term effect of combining suboccipital myofascial release with Maitland mobilization techniques on headache intensity, duration, and frequency, CFRT, upper cervical ROM, general neck mobility, and PPT of upper trapezius and suboccipital muscles.

DETAILED DESCRIPTION:
Cervicogenic headache (CGH) was firstly defined by Ottar Sjaastad a Norwegian neurologist in 1980 as subtype of headache that is irritated by cervical spine movement . CHG is not a primary cause of headache, yet it is a specific type of headache that is caused by different structural abnormalities of the upper neck region leading to neck pain . Headache generally was documented as a high prevalent condition among people. It was classified into three main different types including migraine, tension type and CGH . CGH is common among patients that is responsible for 15-20% of all headache types .

The underlying pathophysiological mechanism of CGH includes any structural abnormality or irritation of the three upper cervical segments (c1, c2 and c3) and muscles supplied by their nerves which consequently led to unilateral referred pain around anatomical bone structures of head, occipital, frontal and temporal regions . Upper cervical pain is the main characteristic of CGH that is presented in 80 percent of the cases . CGH originate from musculoskeletal component disorders such as spine or muscles or disc and another component that aggravates neck pain and mainly arises from upper cervical and atlantooccipital joint that refers symptoms to head or temporal area .

Management of CGH includes pharmacological and non-pharmacological treatment. Regarding the pharmacological treatment, it may relieve pain efficiently, yet, it has many side effects on both short and long term. On the other side, non-pharmacological therapy has positive effects on both pain and function with minimal side effects. It includes manual therapy such as massage, spinal manipulation, and myofascial release, ROM exercises, stretching exercises, strengthening exercise and mobilization techniques aiming at pain relief and curing headache.

The effect of manual therapy had been suggested to be due to modifying sensitivity of the trigeminocervical nucleus . Additionally, myofascial release as a type of manual therapy is observed to relieve pain that is caused by restriction of soft tissue and reduce tissue load that improves eventually ROM (Tavakkoli et al., 2024). Specifically, the myofascial release for the suboccipital region aims at reliving stress and increasing elasticity of suboccipital muscles that were shortened or spasmed due to long and bad body habits such as forward head posture.

The effect of suboccipital release has been documented in different studies according to a systematic review . It improves pain and ROM in patients with CGH. It is used as an immediate pain killer in suboccipital region and improve ROM along cervical and disability of neck during functional activities through correct forward head abnormality.

Another manual therapy technique is Maitland mobilization that includes using oscillation movement at specific joint for enhancing and restoring normal accessory movement of that joint by gliding, rolling, and spinning movement within the joint and is graded according to the aim of treatment . It helps in maintaining normal mobility by normalizing friction between bundle of muscle and nearing structure to reduce pressure on sensitive areas and eventually improving pain and function.

However, there are many authors studied the effect of suboccipital release and the effect of Maitland mobilization on CGH patients, yet, to authors knowledge, there is no study investigated the immediate and short-term combined effect of both suboccipital release with Maitland mobilization. Therefore, this study aims to investigate the immediate and short-term effect of combining suboccipital release with Maitland mobilization on headache intensity, duration, and frequency, cervical flexion rotation test (CFRT), upper cervical ROM, general neck mobility, and pressure pain threshold (PPT) of upper trapezius and suboccipital muscles.

Statement of The Problem This study will be conducted to answer the following question: What is the immediate and short-term effect of combining suboccipital myofascial release with Maitland mobilization techniques on headache intensity, duration, and frequency, CFRT, upper cervical ROM, general neck mobility, and PPT of upper trapezius and suboccipital muscles.

Purpose of The Study This study aims to investigate immediate and short-term effect of combining suboccipital myofascial release with Maitland mobilization techniques on headache intensity, duration, and frequency, CFRT, upper cervical ROM, general neck mobility, and PPT of upper trapezius and suboccipital muscles.

Significance of The Study Headache affects about 66% of population leading to pain, function deterioration, work productivity reduction and increase cost on society. It negatively impacts quality of life .

Suboccipital myofascial release had been documented as an effective method for manging CGH through improve neck disability pain and cervical ROM even than mulligan technique. It is also more effective than conventional physical therapy in reducing pain and intensity of CGH .

On the other hand, Maitland mobilization has been used for a variety of pain and ROM management in mechanical neck pain and CGH. When it had been used combined with postural correction for CGH, it improved pain and function disability more than conventional physical therapy.

As previously mentioned, there are many authors studied the effect of suboccipital release and the effect of Maitland mobilization solely on CGH patients, yet, to authors knowledge, there is no published studies on the immediate nor the short-term effect of combining suboccipital release with Maitland mobilization. Therefore, this study aims to investigate the immediate and short-term effect of combining suboccipital myofascial release with Maitland mobilization on headache intensity, duration, and frequency, CFRT, upper cervical ROM, general neck mobility, and PPT of upper trapezius and suboccipital muscles.

This study will improve the understanding of effective treatments for managing CGH. By examining the combination of soft tissue release with Maitland Mobilization, it highlights how these methods, when used together, can achieve better results in alleviating pain and reducing disability compared to applying each technique individually. This approach targets both joint dysfunction and muscle tension, promoting faster recovery, enhancing quality of life, and lowering healthcare costs. Additionally, this research provides physiotherapists and manual therapists with a practical guide for implementing non-invasive and cost-effective treatment protocols, reducing dependence on pharmacological or surgical interventions. Moreover, this study will broaden the scope for future investigations into combined manual therapy interventions for other musculoskeletal conditions. Ultimately, this study benefits practitioners, patients, and healthcare systems by offering a targeted, interdisciplinary approach to managing CGH effectively.

Delimitation

The study will be delimited to:

* Patients age will range from 20-40 years.
* Fifity- seven patients (both genders) .
* The International Classification of Headache Disorders-III criteria 2018 and CFRT as a base for selecting CGH.
* The VAS for assessing headache intensity.
* The CFRT for diagnosing CGH and evaluating patient progression.
* The CROM device for assessing the upper cervical ROM and the neck general mobility in all directions.
* The pressure algometer for measuring the PPT.

Basic Assumptions

It will be assumed that:

* All patients will follow all the given instructions strictly during the study duration, regarding the assessment and the treatment procedure.
* All participants will be evaluated under the same environmental conditions.

Hypotheses

1. There will be no significant difference between using the three techniques (suboccipital myofascial release alone, Maitland mobilization alone, nor the combined protocol) on headache intensity in patients with CGH neither immediately nor after one week follow up.
2. There will be no significant difference between using the three techniques on headache duration in patients with CGH neither immediately nor after one week follow up.
3. There will be no significant difference between using the three techniques on headache frequency in patients with CGH neither immediately nor after one week follow up.
4. There will be no significant difference between using the three techniques on CFRT in patients with CGH neither immediately nor after one week follow up.
5. There will be no significant difference between using the three techniques on upper cervical ROM in patients with CGH neither immediately nor after one week follow up.
6. There will be no significant difference between using the three techniques on general neck mobility in patients with CGH neither immediately nor after one week follow up.
7. There will be no significant difference between using the three techniques on PPT of upper trapezius muscle in patients with CGH neither immediately nor after one week follow up.
8. There will be no significant difference between using the three techniques on PPT of suboccipital muscle in patients with CGH neither immediately nor after one week follow up.

Definitions of Terms Cervicogenic headache (CGH): It is defined as secondary headache that is associated with cervical disorders and pain originate from upper cervical problem and refer to head and radiate into one or more area and exact mechanism is unknown .

Maitland mobilization: It is one of the popular physical therapy approaches in form of oscillation passive movement of the joint to reduce pain or decrease soft tissue stiffness to increase ROM.

Neck pain: It is a popular musculoskeletal disorder that causes pain in about 67% of people and occurs in upper thoracic spine that physiologically involves movement of neck and shoulder and exacerbate by bad posture.

Pressure pain threshold (PPT): is defined as the minimal amount of pressure where a sense of pressure first changes to pain.

It is defined as nuchal line inhibition technique at muscles surrounding base of the skull and C1 and C2 its technique to release facia by using gentle pressure and stretch for long duration

ELIGIBILITY:
Inclusion Criteria

Each patient will be included in our study if only he/she meets all of the following criteria:

* Age between 20- 40 year.
* No physiotherapy intervention at least for the last three months (Mohamed et al., 2019).
* Neck pain elicited and disturbed by neck movement or maintained position pain produced by pressure over upper cervical (Dunning et al.,2021).
* Limited neck motion with flexion and rotation test less than or equal 32 degree on both right and left side (Dunning et al.,2021).
* Patients suffered from intermittent headaches of varying duration and pain level at least once every week through the last 3 months (Hall et al., 2010; Khalil., et al 2019).

The patient will be excluded if he /she meets one of the following criteria:

* Physical therapy intervention during last three months (Mohamed et al., 2019).
* Primary headaches such as migraine or tension type headache (Mohammadi et al.,2021).
* Cervical radiculopathy, history of neck trauma and previous surgery at neck or shoulder, spondylosis (Mohammadi et al.,2021).
* Vertebrobasilar insufficiency or vestibular dysfunctions (Mohamed et al., 2019).
* Any degenerative vertebral lesion (Shabbir et al., 2021).
* Concomitant medical diagnosis of any primary headache (tension type or migraine) (Shabbir et al., 2021).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
headache intensity | Time Frame: before treatment and one week after treatment
  headache intensity Description: headache intensity which represent the primary outcome by using numerical analogue scale for measure intensity before treatment and one week post treatment

SECONDARY OUTCOMES:
Headache Frequency Headache Duration Cervical Flexion Rotation Test Neck Mobility Assessment Pressure Pain Threshold | Headache Frequency and headache duration before and one week after treatment. Cervical Flexion Rotation Test and Mobility Assessment and Pressure Pain Threshold measurement before and after and one week post treatment
  Headache Frequency number of headache episode per day or week . headache duration time of headache during single episode .Cervical Flexion Rotation Test used for determine. upper cervical lesion Mobility Assessment using CROM device for measure ROM of all neck movement .Pressure Pain Threshold using algometer for measure pain threshold level at suboccipital and upper trapezius muscle

CONTACTS AND LOCATIONS:
Overall Officials: . MAHA MOSTAFA MOHAMMED ALIBEINY, ASS.PROF, Study Director — cairo uneversity faculty of physical therapy
Locations (1):
- Cairo university faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Verma S, Tripathi M, Chandra PS. Cervicogenic Headache: Current Perspectives. Neurol India. 2021 Mar-Apr;69(Supplement):S194-S198. doi: 10.4103/0028-3886.315992. PMID 34003165
- [Result] Priyanka, D. A. T. (2023). A Literature Review to Find the Effectiveness of Suboccipital Myofascial Release Technique in Reducing Cervicogenic Headache. Int J Sci Res, 12(4).
- [Result] Lerner-Lentz A, O'Halloran B, Donaldson M, Cleland JA. Pragmatic application of manipulation versus mobilization to the upper segments of the cervical spine plus exercise for treatment of cervicogenic headache: a randomized clinical trial. J Man Manip Ther. 2021 Oct;29(5):267-275. doi: 10.1080/10669817.2020.1834322. Epub 2020 Nov 5. PMID 33148134